CLINICAL TRIAL: NCT03332212
Title: EMPA-VISION: A Randomised, Double-blind, Placebo-controlled, Mechanistic Cardiac Magnetic Resonance Study to Investigate the Effects of Empagliflozin Treatment on Cardiac Physiology and Metabolism in Patients With Heart Failure
Brief Title: A Study That Looks at the Function of the Heart in Patients With Heart Failure Who Take Empagliflozin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245-0148; 2017-000376-28 (EudraCT Number)
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Empagliflozin + Placebo) (Experimental): Heart Failure with Reduced Ejection Fraction
  Interventions: Drug: Empagliflozin; Drug: Placebo
- Cohort B (Empagliflozin + Placebo) (Experimental): Heart Failure with Preserved Ejection Fraction
  Interventions: Drug: Empagliflozin; Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — 12 weeks
  Other Names: JARDIANCE, JARDIANZ, GIBTULIO
Drug: Placebo — 12 Weeks
  Other Names: JARDIANCE, JARDIANZ, GIBTULIO

SUMMARY:
The objective of this trial is to assess the effect of empagliflozin on cardiac physiology and metabolism aiming to provide a scientific explanation of the underlying mechanism by which empagliflozin improves HF related outcomes in patients with chronic heart failure

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure diagnosed at least 3 months before informed consent
* NYHA class II-IV at screening
* Age ≥ 18 years at screening
* Male or female patients. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Cohort A Heart Failure with Reduced Ejection Fraction (HFrEF)

* Left ventricular ejection fraction (LVEF) ≤ 40% as measured by ECHO at screening
* The following signs of heart failure;

  * Elevated NT-proBNP (>125 pg/mL) at screening in patient without atrial fibrillation (AF)
  * Elevated NT-proBNP (>600 pg/mL) at screening in patient with AF
* Appropriate dose of medical therapy for HF (such as ACEi, ARB, β-blocker, oral diuretics, MRA, ARNI, ivabradine) consistent with prevailing local and international HF guidelines, stable for at least one week prior to Visit 1 and during screening period until Visit 2 (Randomisation) with the exception of diuretics which must be stable for at least one week prior to Visit 2 to control symptoms. If required, the investigator must document in the source documents the reason why the patient is not on the target dose per local guidelines.

Cohort B Heart Failure with Preserved Ejection Fraction (HFpEF)

* Left ventricular ejection fraction (LVEF) ≥ 50% as measured by ECHO at screening and no previous measurement of LVEF ≤ 40%.
* The following combined signs of heart failure;

  * Structural heart disease (LA enlargement [LAVI >34 mL/m2] and/or LVH [LVMI ≥ 115 g/m2 for males and ≥ 95 g/m2 for females]) by ECHO at screening or within 3 months prior to informed consent AND
  * NT-proBNP > 125pg/mL at screening in patient without AF or NT-pro-BNP > 600 pg/mL in patient with AF
* Oral diuretics, if prescribed, should be stable for at least one week prior to Visit 1 and during screening period until Visit 2 (Randomisation).

Exclusion Criteria:

* Stroke or transient ischaemic attack (TIA) within 6 months prior to informed consent.
* Any patients with myocardial scars and/or non-viable myocardium in the interventricular septum, unstable angina due to significant coronary artery disease (CAD), or major (in the opinion of the investigator) cardiovascular surgery.
* Any contraindication for MRI, CPET and/or dobutamine stress test in accordance with the institution guidance, including implanted left ventricular assist device (LVAD),implantable cardioverter defibrillator (ICD), cardiac resynchronisation therapy (CRT) or any cardiac device.
* Heart transplant recipient or listed for heart transplant
* Cardiomyopathy based on infiltrative diseases (e.g. amyloidosis), accumulation diseases (e.g. haemochromatosis, Fabry disease), muscular dystrophies, cardiomyopathy with reversible causes (e.g. stress cardiomyopathy), hypertrophic obstructive cardiomyopathy or known pericardial constriction
* Moderate to severe uncorrected valvular heart disease, obstructive or regurgitant, or any valvular heart disease expected to lead to surgery in the Investigator's opinion
* Acute decompensated HF (exacerbation of chronic HF) requiring intravenous (i.v.) diuretics, i.v. inotropes or i.v. vasodilators, or LVAD or hospitalisation within 1 week prior to Visit 1 (Screening), or during screening period until Visit 2 (Randomisation)
* Systolic blood pressure (SBP) ≥ 180 mmHg at screening. If SBP >150 mmHg and <180mmHg at screening, the patient is ineligible if receiving 3 or more antihypertensive drugs
* Symptomatic hypotension and/or a SBP < 100 mmHg at Screening
* Atrial fibrillation which is uncontrolled in the opinion of the investigator
* Untreated ventricular arrhythmia with syncope documented within the 3 months prior to informed consent in patients without ICD
* Diagnosis of cardiomyopathy induced by chemotherapy or peripartum within the 12 months prior to informed consent
* Symptomatic bradycardia or second or third degree heart block in need of a pacemaker after adjusting beta-blocker therapy or any other negative inotropic agents, if appropriate
* Chronic pulmonary disease requiring home oxygen, oral steroid therapy or hospitalisation for exacerbation within 12 months prior to informed consent, or significant chronic pulmonary disease in the Investigator's opinion, or primary pulmonary arterial hypertension
* Indication of liver disease, defined by serum levels of either ALT (SGPT), AST (SGOT),or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined at screening
* Impaired renal function, defined as estimated Creatinine Clearance < 30 mL/min (using Cockcroft-Gault formula) or requiring dialysis, as determined at screening
* Haemoglobin < 10 g/dL at screening
* Type 1 Diabetes Mellitus (T1DM)
* History of ketoacidosis
* Major surgery (major according to the investigator's assessment) performed within 3 months prior to informed consent, or scheduled major elective surgery (e.g. hip replacement) within 3 months after Visit 1
* Gastrointestinal (GI) surgery or GI disorder that could interfere with absorption of trial medication in the investigator's opinion
* Any documented active or suspected malignancy or history of malignancy within 6 months prior to informed consent, except appropriately treated basal cell carcinoma of the skin, in situ carcinoma of uterine cervix or low risk prostate cancer (patients with pretreatment PSA <10 ng/mL, and biopsy Gleason score of ≤ 6 and clinical stage T1c or T2a)
* Presence of any other disease than heart failure with a life expectancy of <1 year in the investigator's opinion
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Patients with requirement for treatment with empagliflozin according to local standard of care
* Treatment with any SGLT-2 inhibitor or combined SGLT-1 and 2 inhibitor within 1 week prior to informed consent or during screening period until Visit 2 (Randomisation)
* Currently enrolled in another investigational device or drug study, or less than 30 days between randomisation and ending another investigational device or drug study, or receiving other investigational treatment(s). Patients participating in a purely observational trial will not be excluded.
* Known allergy or hypersensitivity to empagliflozin or other SGLT-2 inhibitors
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable trial subject or unlikely to complete the trial
* Women who are pregnant, breastfeeding, or who plan to become pregnant while in the trial
* Any clinical condition that would jeopardise patients safety while participating in this trial, or may prevent the subject from adhering to the trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] Hundertmark MJ, Adler A, Antoniades C, Coleman R, Griffin JL, Holman RR, Lamlum H, Lee J, Massey D, Miller JJJJ, Milton JE, Monga S, Mozes FE, Nazeer A, Raman B, Rider O, Rodgers CT, Valkovic L, Wicks E, Mahmod M, Neubauer S. Assessment of Cardiac Energy Metabolism, Function, and Physiology in Patients With Heart Failure Taking Empagliflozin: The Randomized, Controlled EMPA-VISION Trial. Circulation. 2023 May 30;147(22):1654-1669. doi: 10.1161/CIRCULATIONAHA.122.062021. Epub 2023 Apr 18. PMID 37070436
- [Derived] Hundertmark MJ, Agbaje OF, Coleman R, George JT, Grempler R, Holman RR, Lamlum H, Lee J, Milton JE, Niessen HG, Rider O, Rodgers CT, Valkovic L, Wicks E, Mahmod M, Neubauer S. Design and rationale of the EMPA-VISION trial: investigating the metabolic effects of empagliflozin in patients with heart failure. ESC Heart Fail. 2021 Aug;8(4):2580-2590. doi: 10.1002/ehf2.13406. Epub 2021 May 6. PMID 33960149
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomised, double-blind, placebo controlled, mechanistic cardiac magnetic resonance study to investigate the effects of empagliflozin treatment on cardiac physiology and metabolism in patients with heart failure.
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist site to ensure that they (the subjects) met all implemented inclusion/exclusion criteria.
Groups:
- Placebo Cohort A: Once a day oral administration of a single film-coated placebo tablet matching to empagliflozin for 12 weeks.
  Cohort A: Heart failure (HF) with reduced ejection fraction (HFrEF).
- Placebo Cohort B: Once a day oral administration of a single film-coated placebo tablet matching to empagliflozin for 12 weeks.
  Cohort B: Heart failure (HF) with preserved ejection fraction (HFpEF).
- Empagliflozin 10mg Cohort A: Once a day oral administration of a single 10 milligram (mg) film-coated empagliflozin tablet for 12 weeks.
  Cohort A: Heart failure (HF) with reduced ejection fraction (HFrEF).
- Empagliflozin 10mg Cohort B: Once a day oral administration of a single 10 milligram (mg) film-coated empagliflozin tablet for 12 weeks.
  Cohort B: Heart failure (HF) with preserved ejection fraction (HFpEF).
Period: Overall Study
Arm/Group | Placebo Cohort A | Placebo Cohort B | Empagliflozin 10mg Cohort A | Empagliflozin 10mg Cohort B
Started | 19 | 18 | 17 | 18
Treated | 19 | 17 | 17 | 18
Completed | 18 | 16 | 17 | 17
Not Completed | 1 | 2 | 0 | 1
Not completed — Not treated | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — worsening of disease under study | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomised set (RS): This set included all patients who were randomised to study treatment, in line with the intention-to-treat principle.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Cohort A | Placebo Cohort B | Empagliflozin 10mg Cohort A | Empagliflozin 10mg Cohort B | Total
Number analyzed (Participants) | 19 | 18 | 17 | 18 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (12.7) | 72.1 (7.0) | 67.5 (14.1) | 69.1 (10.9) | 68.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 7 | 8 | 30
  Male | 13 | 9 | 10 | 10 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 18 | 17 | 18 | 72
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 19 | 18 | 17 | 16 | 70
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ratio of phosphocreatine to adenosine triphosphate concentration [Mean (Standard Deviation); unit: Ratio] — The ratio of phosphocreatine to adenosine triphosphate concentration (PCr/ATP) reflects the energetic state of the heart and was assessed by 31P cardiac magnetic resonance spectroscopy (MRS). Population: In the Placebo arm (Cohort B) there was one patient without baseline Cardiac magnetic resonance (CMR) measures.
  Ratio
    number analyzed (Participants) | 19 | 17 | 17 | 18 | 71
    (all) | 1.924 (0.354) | 1.719 (0.431) | 1.889 (0.407) | 1.896 (0.462) | 1.859 (0.413)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in PCr/ATP Ratio in the Resting State Measured by 31P Cardiac Magnetic Resonance Spectroscopy (MRS).
Description: The primary endpoint of efficacy was the change from baseline to Week 12 in phosphocreatine/adenosine triphosphate (PCr/ATP) ratio in the resting state measured by 31P cardiac magnetic resonance spectroscopy (MRS).
  Adjusted mean values were calculated using an analysis of variance (ANOVA) model, with treatment, history of diabetes, and history of atrial fibrillation (AF) as fixed effects.
Time Frame: At baseline and at week 12.
Population: Per protocol set (PPS):
  The primary endpoint analysis was performed using the per protocol (PP) set of patients with valid PCr/ATP ratio measurements available at baseline and Week 12, and no important protocol violation relevant to the primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: PCr / ATP Ratio
Arm/Group | Placebo Cohort A | Placebo Cohort B | Empagliflozin 10mg Cohort A | Empagliflozin 10mg Cohort B
Number analyzed (Participants) | 18 | 11 | 17 | 13
PCr / ATP Ratio | 0.068 (0.114) | 0.259 (0.156) | -0.179 (0.117) | 0.100 (0.143)
Statistical Analysis 1: Comparison: Placebo Cohort A vs Empagliflozin 10mg Cohort A; ANOVA on the PCr/ATP ratio absolute change using treatment (empagliflozin vs. placebo), history of diabetes (yes vs, no) and history of atrial fibrillation (yes vs no) as between subjects factor; Test type: Other; p = 0.1418, ANOVA; Mean Difference (Final Values) = -0.247, 95% CI 2-sided [-0.582 to 0.087], Standard Error of Mean 0.164
Statistical Analysis 2: Comparison: Placebo Cohort B vs Empagliflozin 10mg Cohort B; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.4650, ANOVA; Mean Difference (Final Values) = -0.159, 95% CI 2-sided [-0.604 to 0.286], Standard Error of Mean 0.213

ADVERSE EVENTS:
Time Frame: All adverse events occurring between the start of treatment and end of the residual effect period, 7 days after the last dose of medication. Up to 95 days.
Description: Treated set (TS): All randomised and treated patients were included in the safety analysis and safety summaries were presented by actual treatment received.
Groups:
- Placebo: Once a day oral administration of a single film-coated placebo tablet matching to empagliflozin for 12 weeks. Cohort A: Heart failure (HF) with reduced ejection fraction (HFrEF) and Cohort B: Heart failure (HF) with preserved ejection fraction (HFpEF).
- Empagliflozin 10mg: Once a day oral administration of a single 10 milligram (mg) film-coated empagliflozin tablet for 12 weeks. Cohort A: Heart failure (HF) with reduced ejection fraction (HFrEF) and Cohort B: Heart failure (HF) with preserved ejection fraction (HFpEF).
Arm/Group | Placebo | Empagliflozin 10mg
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 7/36 | 1/35
Other Adverse Events (participants affected / at risk) | 3/36 | 8/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | Empagliflozin 10mg (N=35)
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Glaucoma (Eye disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Euglycaemic diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=36) | Empagliflozin 10mg (N=35)
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Due to the suspension of face-to-face contact imposed in March 2020 to restrict transmission of COVID-19, the number of patients included in the analysis of efficacy for the Heart failure with preserved ejection fraction was substantially reduced, which meant that this cohort was also under powered (reduced from 80% to 70%) for the planned analysis of the primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT03332212/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT03332212/SAP_001.pdf